CLINICAL TRIAL: NCT06509204
Title: Real-world Evaluation of JBA GlucoTrojan With Reducose® on Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tastermonial Inc (Industry)
Collaborators: WCG clinical (Unknown); Affordable Quality Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1351713
Record Dates: First submitted 2024-06-28; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Food Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consumer (Experimental): AQP Pharmaceuticals, Inc. ("Company") developed a powdered supplement sachet that can be added to meals targeting consumers who follow carbohydrate-heavy Asian diets. The product is formulated with the patented ingredient, "Reducose®", a natural water extract of novel White Mulberry Leaf that has been scientifically proven to reduce the absorption of sugars and other carbs by up to 40%. The effects have been confirmed previously via Randomized, Double-Blind, Controlled Trials.
  The Company is looking to conduct a real-world study of blood glucose responses to JBA GlucoTrojan (see specifications here) with a 5% concentration of Reducose®. The study will observe the real-world efficacy of GlucoTrojan when taken with high carbohydrate meals.
  Interventions: Dietary Supplement: Glucotrojan

INTERVENTIONS:
Dietary Supplement: Glucotrojan — Day 1: Start wearing the CGM sensor and let it self-calibrate for 24 h Day 2: Consume 1 serving of Test Meal for breakfast. Log the meal in the app. Day 3: Consume 1 serving of Test Meal with GlucoTrojan for breakfast. Log the meal in the app.
  Days 4-8: Participants will be instructed to take GlucoTrojan twice per day. Once during their typical breakfast meal and once during their typical dinner meal. Each breakfast and dinner will be logged in the app.
  Days 9-13: Participants will continue with their typical lives but continue to log meals - breakfast and dinner - in the app.
  Day 14: end

SUMMARY:
The project is focused on evaluating the real-world efficacy of JBA GlucoTrojan, a powdered supplement sachet containing Reducose, a natural water extract of White Mulberry Leaf, which has been scientifically proven to reduce the absorption of sugars and carbs by up to 40%. The study aims to compare the effect of consuming GlucoTrojan with a meal (Test Meal) vs. having the meal alone (control) on the blood sugar response of 50 healthy adults, pre-diabetes, or non-insulin dependent diabetes, over a period of 14 days. It is expected that GlucoTrojan will reduce the incremental area under the curve and the peak for plasma glucose concentration over 120 minutes in normoglycemic adults when compared to the response to a control meal.

ELIGIBILITY:
Inclusion criteria:

* Consent to study protocol
* BMI: 18.5 to 29.9 kg/m2
* 21 to 75 years old

Exclusion criteria:

* Physician-diagnosed T1D and insulin-dependent T2D
* Taking medications that modulate blood glucose response or control blood pressure other than Metformin
* An underlying health condition that warrants non-participation
* Individuals who are pregnant
* Any other dietary restrictions that prevent them from consuming study foods
* Unable to follow remote guidance via the Internet or smartphone
* Unable to follow controlled diet instructions
* Unable to use a CGM (Continuous Glucose Monitoring Devices)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
iAUC Calculation | 2-hour period after eating
  Each participant's eating period (called a "meal") is normalized and overlaid in a data frame that captures glucose values over the course of the test. Several other metrics are computed, such as maximum and minimum values, standard deviation, and others. In particular, the iAUC ("incremental area under the curve"), a measure of the total amount of postprandial blood glucose level increased over the entire 2-hour period after eating. The methodology of iAUC calculation follows the gold standard used in the measurement of the glycemic index (1, 2). The iAUC metric allows our team to easily compare and rank testing results, as well as compare against the pure sugar responses or the sugar tolerance test of an individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Tastermonial, Cupertino, California, United States

REFERENCES:
- [Background] Freckmann G, Hagenlocher S, Baumstark A, Jendrike N, Gillen RC, Rossner K, Haug C. Continuous glucose profiles in healthy subjects under everyday life conditions and after different meals. J Diabetes Sci Technol. 2007 Sep;1(5):695-703. doi: 10.1177/193229680700100513. PMID 19885137
- [Background] Zhou J, Li H, Ran X, Yang W, Li Q, Peng Y, Li Y, Gao X, Luan X, Wang W, Jia W. Reference values for continuous glucose monitoring in Chinese subjects. Diabetes Care. 2009 Jul;32(7):1188-93. doi: 10.2337/dc09-0076. Epub 2009 Apr 23. PMID 19389816
- [Background] Shah VN, DuBose SN, Li Z, Beck RW, Peters AL, Weinstock RS, Kruger D, Tansey M, Sparling D, Woerner S, Vendrame F, Bergenstal R, Tamborlane WV, Watson SE, Sherr J. Continuous Glucose Monitoring Profiles in Healthy Nondiabetic Participants: A Multicenter Prospective Study. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4356-4364. doi: 10.1210/jc.2018-02763. Erratum In: J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1775-e1776. doi: 10.1210/clinem/dgab837. PMID 31127824
- [Background] Rodriguez-Segade S, Rodriguez J, Camina F, Fernandez-Arean M, Garcia-Ciudad V, Pazos-Couselo M, Garcia-Lopez JM, Alonso-Sampedro M, Gonzalez-Quintela A, Gude F. Continuous glucose monitoring is more sensitive than HbA1c and fasting glucose in detecting dysglycaemia in a Spanish population without diabetes. Diabetes Res Clin Pract. 2018 Aug;142:100-109. doi: 10.1016/j.diabres.2018.05.026. Epub 2018 May 26. PMID 29807103
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Fox LA, Beck RW, Xing D. Variation of interstitial glucose measurements assessed by continuous glucose monitors in healthy, nondiabetic individuals. Diabetes Care. 2010 Jun;33(6):1297-9. doi: 10.2337/dc09-1971. Epub 2010 Mar 9. PMID 20215454

DOCUMENTS (1):
  • Study Protocol (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT06509204/Prot_000.pdf